CLINICAL TRIAL: NCT07139847
Title: Effect of Intraoperative Magnesium Infusion on Postoperative Emergence Agitation in Patients Undergoing Lumbar Microdiscectomy
Brief Title: Magnesium Sulfate for Prevention of Emergence Agitation in Lumbar Disc Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, M.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GUAH-MAG-2025-01
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Disc Herniation; Emergence Agitation; Magnesium Sulfate
Keywords: Magnesium Sulfate; Lumbar Disc Herniation; Postoperative Complications
MeSH Terms: conditions — Intervertebral Disc Displacement; Emergence Delirium; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups: the experimental group receiving intraoperative magnesium sulfate infusion and the control group receiving an equivalent volume of 0.9% saline. Both groups will be managed under a standardized general anesthesia protocol, and outcomes will be assessed in the post-anesthesia care unit (PACU) by blinded evaluators.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both participants and clinical staff (including anesthesia providers) were blinded to group allocation. Group assignments were determined using sealed opaque envelopes and were only known to an anesthesia technician not involved in patient care or outcome assessment. The infusion solutions (magnesium sulfate or 0.9% saline) were prepared in identical syringes to maintain blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate Infusion (Active Comparator): Participants assigned to this group will receive an intravenous bolus of magnesium sulfate 30 mg/kg over 15 minutes immediately after induction of general anesthesia, followed by continuous infusion at 10 mg/kg/h until the end of surgery.
  Interventions: Drug: Magnesium Sulfate Infusion
- 0.9% Saline Infusion (Placebo Comparator): Participants assigned to this group will receive an intravenous bolus and continuous infusion of 0.9% sodium chloride solution in the same volume, infusion rate, and duration as the magnesium sulfate group
  Interventions: Drug: 0.9% Saline Infusion

INTERVENTIONS:
Drug: Magnesium Sulfate Infusion — Magnesium Sulfate (Experimental Group) Intravenous bolus of magnesium sulfate 30 mg/kg administered over 15 minutes immediately after induction of general anesthesia, followed by continuous infusion at 10 mg/kg/h until the end of surgery. Solutions were prepared in identical syringes and infusion bags by an anesthesia technician not involved in patient care. The preparation and administration protocol ensured blinding of participants, anesthesia providers, and outcome assessors.
  Arms: Magnesium Sulfate Infusion
Drug: 0.9% Saline Infusion — ntravenous bolus and continuous infusion of 0.9% sodium chloride solution in the same volume, infusion rate, and duration as the magnesium sulfate group. Solutions were indistinguishable in appearance and prepared under the same blinding procedures.
  Arms: 0.9% Saline Infusion

SUMMARY:
This randomized, double-blind, controlled trial investigates the effect of intraoperative magnesium sulfate infusion on the incidence of postoperative emergence agitation in adult patients undergoing elective lumbar microdiscectomy under general anesthesia. Eligible participants (ASA physical status I-II, aged 18-70 years) will be randomly assigned to receive either magnesium sulfate or 0.9% saline during surgery. The primary outcome is the incidence of emergence agitation in the post-anesthesia care unit (PACU), assessed at admission and at 5, 10, 15, and 30 minutes using the Ramsay Sedation Scale. Secondary outcomes include postoperative pain scores (Numeric Rating Scale), intraoperative remifentanil consumption, recovery and extubation times, tramadol use in the PACU, and any adverse events related to magnesium infusion.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, controlled trial will be conducted at Ondokuz Mayis University and Giresun Training and Research Hospital. The study aims to evaluate the effect of intraoperative magnesium sulfate infusion on postoperative emergence agitation (EA) in patients undergoing elective lumbar microdiscectomy under general anesthesia.

Following ethics committee approval and written informed consent, adult patients aged 18-70 years, classified as ASA physical status I or II, scheduled for single-level lumbar microdiscectomy, will be enrolled. Exclusion criteria include severe cardiovascular disease, psychiatric disorders, neuromuscular disease, pregnancy, hepatic or renal dysfunction, use of calcium channel blockers, hypnotics, anxiolytics, antipsychotics, allergy to study drugs, or refusal to participate.

Participants will be randomized (1:1) using a computer-generated sequence to either:

Magnesium Group (Group M): 30 mg/kg magnesium sulfate IV bolus over 15 minutes after induction, followed by continuous infusion at 10 mg/kg/h until the end of surgery.

Control Group (Group K): Equivalent volume and rate of 0.9% saline.

All patients will receive standardized anesthesia, including premedication with midazolam, induction with propofol, fentanyl, and rocuronium, and maintenance with sevoflurane in 50% air/oxygen mixture. Remifentanil infusion (0.1-0.25 µg/kg/min) will be adjusted to maintain target bispectral index (BIS) values between 40 and 60.

The primary outcome is the incidence of emergence agitation in the post-anesthesia care unit (PACU), measured at admission (T0) and at 5 (T1), 10 (T2), 15 (T3), and 30 (T4) minutes post-admission using the Ramsay Sedation Scale (RSS).

Secondary outcomes include Numeric Rating Scale (NRS) pain scores at the same PACU time points, total intraoperative remifentanil consumption, recovery time (from sevoflurane discontinuation to eye opening), extubation time (from sevoflurane discontinuation to extubation), meperidine use in the PACU, and the incidence of adverse events (arrhythmia, neuromuscular blockade, respiratory difficulties) related to magnesium infusion.

Sample size was calculated based on pilot data, requiring 32 participants per group for 80% power at a 0.05 significance level, with 35 enrolled per group to account for potential dropouts. Statistical analysis will use Student's t-test or Mann-Whitney U test for continuous variables, Chi-square or Fisher's exact test for categorical variables, with significance set at p < 0.05. Analyses will be performed using SPSS v25.0.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 70 years

ASA physical status classification I or II

Scheduled for elective single-level lumbar microdiscectomy under general anesthesia

Ability to provide written informed consent

Exclusion Criteria:

Severe cardiovascular disease

History of psychiatric disorder

Neuromuscular disease

Pregnancy or breastfeeding

Hepatic or renal dysfunction

Current use of calcium channel blockers, hypnotics, anxiolytics, or antipsychotic medications

Known allergy to magnesium sulfate or study-related medications

Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Agitation in the PACU | At PACU admission (T0) and at 5, 10, 15, and 30 minutes post-admission.
  Percentage of participants with a Ramsay Sedation Scale (RSS) score ≥5, indicating emergence agitation, in the post-anesthesia care unit (PACU)

SECONDARY OUTCOMES:
Postoperative Pain Scores in PACU | At PACU admission (T0) and at 5, 10, 15, and 30 minutes post-admission.
  Numeric Rating Scale (NRS) pain scores ranging from 0 (no pain) to 10 (worst pain).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and institutional policies.

REFERENCES:
- [Result] 1. McKeown, A., & Agarwala, R. (2020). "Emergence agitation: Recognition, prevention, and treatment." BJA Education, 20(6), 180-184. https://doi.org/10.1016/j.bjae.2020.03.002
- [Result] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Result] Soltész, P., Silvasti, M., & Taivainen, T. (2013). "Emergence agitation in adults after general anesthesia: A comparison of sevoflurane and propofol." Acta Anaesthesiologica Scandinavica, 57(3), 315-321. https://doi.org/10.1111/aas.12047